CLINICAL TRIAL: NCT02028260
Title: Modafinil vs. Placebo for Hypoactive Delirium in the Critically Ill: A Randomized, Controlled Trial
Brief Title: Modafinil Versus Placebo for Hypoactive Delirium in the Critically Ill
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: unable to enroll
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Gerald L. Weinhouse, BWPO PHYSICIAN, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013P002105
Record Dates: First submitted 2013-12-19; First posted 2014-01-07 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Delirium; Respiratory Failure
MeSH Terms: conditions — Delirium; Respiratory Insufficiency | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Modafinil (Active Comparator): Modafinil 200 mg qAM enterally for the duration the patient is confirmed to be in a hypoactive delirium to a maximum of 14 days.
  Interventions: Drug: Modafinil
- Placebo (Placebo Comparator): normal saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Modafinil — 200 mg daily
  Other Names: provigil
  Arms: Modafinil
Drug: Placebo — similar appearing inert tablet
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo controlled study of 30 patients. Patients who qualify, as per the inclusion criteria (RASS greater than -3, less then +1, CAM positive, present gastric access) will either be given 200mg of modafinil or an identical, indistinguishable placebo. The placebo and study drug will be distributed by the hospital pharmacy. Once enrolled, each patient will be reassessed every morning to determine appropriateness for drug administration. If the RASS is less than -3 (i.e. comatose) or greater then 0 modafinil will not be given. He/she will then be assessed each morning thereafter. Due to the stimulant-like actions of modafinil, the drug will be administered only in the morning. Patients will be assessed for delirium at least twice a day; trained personnel using the Confusion Assessment Method (CAM) will do the assessment. Qualification for a delirium free day will be no positive CAM screens for 24 hours following drug administration. Additional data such as days on mechanical ventilation and progression to tracheotomy will also be collected hypothesizing that patients who take modafinil will have a shorter time to extubation therefore avoiding the need for a tracheotomy. Post-discharge from the unit, but within 48 hours, patients will be asked to participate in a survey (The Richards-Campbell Sleep Questionnaire (RCSQ) assessing their perception of daytime and nighttime sleepiness in the intensive care unit as well as their overall perception of rest. Their functional capacity will also be evaluated at this time and compared to their pre-morbid baseline. The hypothesis tested is that Modafinil restores sleep cycle synchrony in the ICU therefore increasing delirium free days and improving ICU outcomes.

DETAILED DESCRIPTION:
Eligibility Criteria

Inclusion Criteria To be eligible for study entry, subjects must satisfy these main criteria

Inclusion criteria:

3.1 Inclusion Criteria

* Adult patients ≥ 18 yrs of age, < 76 yrs of age
* Admitted to MICU (3B and 3C) or SICU (8C, 8D, 11C)
* Surrogate present to provide informed consent when patient is not able
* RASS score of >-3, < +1
* CAM positive
* Enteral access

3.2 Exclusion Criteria:

* Recent MI (within past 2 weeks)
* High risk of dysrhythmias (i.e. bundle branch block, QT prolongation, class IV HF, implanted device)
* Unable to tolerate enteral medication
* History of stimulant induced mania/psychosis
* Pre-existing neurologic disease
* Patients transferred from outside hospital
* Pregnancy
* Alcohol withdrawal
* History of end stage liver disease (Childs-Pugh class B or worse)
* Prognosis considered hopeless (CMO)

ELIGIBILITY:
Inclusion Criteria

* Adult patients ≥ 18 yrs of age, < 76 yrs of age
* Admitted to MICU (3B and 3C) or SICU (8C, 8D, 11C)
* Surrogate present to provide informed consent when patient is not able
* RASS score of >-3, < +1
* CAM positive
* Enteral access

Exclusion Criteria:

* Recent MI (within past 2 weeks)
* High risk of dysrhythmias (i.e. bundle branch block, QT prolongation, class IV HF, implanted device)
* Unable to tolerate enteric medication
* History of stimulant induced mania/psychosis
* Pre-existing neurologic disease
* Patients transferred from outside hospital
* Pregnancy
* Alcohol withdrawal
* History of end stage liver disease (Childs-Pugh class B or worse)
* Prognosis considered hopeless (CMO)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2015-07 (Estimated); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Decreased CAM positive days in the ICU | Up to 14 days of ICU stay

SECONDARY OUTCOMES:
Length of stay in the ICU | Up to 14 days of ICU stay

OTHER OUTCOMES:
Patients perception of their sleep pattern in the ICU | Up to 14 days of ICU stay
Return to baseline activities of daily living (ADL's) | Up to 14 days of ICU stay
Amount of psychotropic medication co-administered | Up to 14 days of ICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Gerald L Weinhouse, MD, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts